CLINICAL TRIAL: NCT04513717
Title: Parallel Phase III Randomized Trials for High Risk Prostate Cancer Evaluating De-Intensification for Lower Genomic Risk and Intensification of Concurrent Therapy for Higher Genomic Risk With Radiation (PREDICT-RT*)
Brief Title: Two Studies for Patients With High Risk Prostate Cancer Testing Less Intense Treatment for Patients With a Low Gene Risk Score and Testing a More Intense Treatment for Patients With a High Gene Risk Score, The PREDICT-RT Trial
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU009; NCI-2020-04705 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU009 (Other: NRG Oncology); NRG-GU009 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2020-08-07; First posted 2020-08-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma; Stage III Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; bicalutamide; Specimen Handling; Buserelin; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Flutamide; Salicylic Acid; Goserelin; histrelin; Leuprolide; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; relugolix; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (de-intensification study) (Active Comparator): Patients undergo RT over 2-11 weeks and receive ADT (consisting of either leuprolide, goserelin, triptorelin, degarelix, buserelin, histrelin, or relugolix and bicalutamide or flutamide) for 24 months in the absence of disease progression or unacceptable toxicity. Patients undergo bone scan, PET scan, CT scan, and MRI at screening and as clinically indicated and may optionally undergo blood sample collection throughout the study.
  Interventions: Drug: Bicalutamide; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Buserelin; Procedure: Computed Tomography; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin; Drug: Histrelin; Drug: Leuprolide; Procedure: Magnetic Resonance Elastography; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Relugolix; Drug: Triptorelin
- Arm II (de-intensification study) (Experimental): Patients undergo RT over 2-11 weeks and receive ADT (consisting of either leuprolide, goserelin, triptorelin, degarelix, buserelin, histrelin, or relugolix and bicalutamide or flutamide) for 12 months in the absence of disease progression or unacceptable toxicity. Patients undergo bone scan, PET scan, CT scan, and MRI at screening and as clinically indicated and may optionally undergo blood sample collection throughout the study.
  Interventions: Drug: Bicalutamide; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Buserelin; Procedure: Computed Tomography; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin; Drug: Histrelin; Drug: Leuprolide; Procedure: Magnetic Resonance Elastography; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Relugolix; Drug: Triptorelin
- Arm III (intensification study) (Active Comparator): Patients undergo RT over 2-11 weeks and receive ADT as in Arm I. Patients undergo bone scan, PET scan, CT scan, and MRI at screening and as clinically indicated and may optionally undergo blood sample collection throughout the study.
  Interventions: Drug: Bicalutamide; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Buserelin; Procedure: Computed Tomography; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin; Drug: Histrelin; Drug: Leuprolide; Procedure: Magnetic Resonance Elastography; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Relugolix; Drug: Triptorelin
- Arm IV (intensification study) (Experimental): Patients undergo RT over 2-11 weeks and receive ADT (consisting of either leuprolide, goserelin, triptorelin, degarelix, buserelin, histrelin, or relugolix) for 24 months in the absence of disease progression or unacceptable toxicity. Patients also receive apalutamide PO QD. Treatment repeats every 90 days for up to 8 cycles (24 months) in the absence of disease progression or unacceptable toxicity. Patients undergo bone scan, PET scan, CT scan, and MRI at screening and as clinically indicated and may optionally undergo blood sample collection throughout the study.
  Interventions: Drug: Apalutamide; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Buserelin; Procedure: Computed Tomography; Drug: Degarelix; Drug: Goserelin; Drug: Histrelin; Drug: Leuprolide; Procedure: Magnetic Resonance Elastography; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Relugolix; Drug: Triptorelin

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
  Arms: Arm IV (intensification study)
Drug: Bicalutamide — Given bicalutamide
  Other Names: Casodex; Cassotide; Cosudex; ICI 176,334; ICI 176334; Utamide
  Arms: Arm I (de-intensification study); Arm II (de-intensification study); Arm III (intensification study)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Buserelin — Given buserelin
  Other Names: 6-[O-(1,1-Dimethylethyl)-D-serine]-9-(N-ethyl-L-prolinamide)-10-deglycinamide-luteinizing Hormone-releasing Factor (Pig); BSRL; Busereline; Etilamide; HOE 766; HOE-766; HOE766; ICI 123215; ICI-123215; ICI123215; S74 6766; S74-6766; S746766; Tiloryth
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Degarelix — Given degarelix
  Other Names: ASP 3550; ASP-3550; ASP3550; FE 200486; FE-200486; FE200486; Firmagon
Drug: Flutamide — Given flutamide
  Other Names: 4'-Nitro-3'-trifluoromethylisobutyranilide; Apimid; Cebatrol; Chimax; Cytomid; Drogenil; Euflex; Eulexine; Flucinom; Flucinome; Flugerel; Fluken; Flulem; FLUT; Fluta-Gry; Flutabene; Flutacan; Flutamex; Flutamin; Flutan; Flutaplex; Fugerel; Grisetin; Niftolide; Oncosal; Profamid; Propanamide, 2-Methyl-N-(4-nitro-3-(trifluoromethyl)phenyl)-; Prostacur; Prostadirex; Prostica; Prostogenat; Sch 13521; Tafenil; Tecnoflut; Testotard
  Arms: Arm I (de-intensification study); Arm II (de-intensification study); Arm III (intensification study)
Drug: Goserelin — Given goserelin
  Other Names: ICI-118630
Drug: Histrelin — Given histrelin
Drug: Leuprolide — Given leuprolide
  Other Names: Leuprorelin
Procedure: Magnetic Resonance Elastography — Undergo MRI
  Other Names: MRE
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Relugolix — Given relugolix
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; Relumina; TAK 385; TAK-385; TAK385
Drug: Triptorelin — Given triptorelin
  Other Names: 6-D-Tryptophan-LH-RH; 6-D-Tryptophanluteinizing Hormone-releasing Factor; AY 25650; AY-25650; AY25650; CL 118532; CL-118,532; CL-118532; CL118532; Detryptoreline

SUMMARY:
This phase III trial compares less intense hormone therapy and radiation therapy to usual hormone therapy and radiation therapy in treating patients with high risk prostate cancer and low gene risk score. This trial also compares more intense hormone therapy and radiation therapy to usual hormone therapy and radiation therapy in patients with high risk prostate cancer and high gene risk score. Apalutamide may help fight prostate cancer by blocking the use of androgen by the tumor cells. Radiation therapy uses high energy rays to kill tumor cells and shrink tumors. Giving a shorter hormone therapy treatment may work the same at controlling prostate cancer compared to the usual 24 month hormone therapy treatment in patients with low gene risk score. Adding apalutamide to the usual treatment may increase the length of time without prostate cancer spreading as compared to the usual treatment in patients with high gene risk score.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether men with National Comprehensive Cancer Network (NCCN) high risk prostate cancer who are in the lower 2/3 of Decipher genomic risk (=< 0.85) can be treated with 12 months androgen deprivation therapy (ADT) plus radiation therapy (RT) instead of 24 months ADT+RT and experience non-inferior metastasis-free survival. (De-intensification study) II. To determine whether men with NCCN high risk prostate cancer who are in the upper 1/3 of Decipher genomic risk (> 0.85) or have node-positive disease by conventional imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) will have a superior metastasis-free survival (MFS) through treatment intensification with apalutamide added to the standard of RT plus 24 month ADT. (Intensification study)

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) between the standard of care (RT plus 24 months of ADT) and either the de-intensification (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies) II. To compare time to prostate specific antigen (PSA) failure or start of salvage treatment between the standard of care (RT plus 24 months of ADT) and either the de-intensification arm (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies) III. To compare PSA failure-free survival with non-castrate testosterone and no additional therapies between the standard of care (RT plus 24 months of ADT) and either the de-intensification arm (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies) IV. To compare MFS judged based on either standard or molecular imaging between the standard of care (RT plus 24 months of ADT) and either the de-intensification arm (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies) V. To compare prostate cancer-specific mortality between the standard of care (RT plus 24 months of ADT) and either the de-intensification arm (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies) VI. To compare testosterone levels at the time of PSA failure and metastases between the standard of care (RT plus 24 months of ADT) and either the de-intensification arm (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies) VII. To compare time to testosterone recovery (defined as a T > 200) between the standard of care (RT plus 24 months of ADT) and either the de-intensification arm (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies) VIII. To compare adverse events, both clinician-reported using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 and patient-reported using Patient Reported Outcome (PRO)-CTCAE items, between the standard of care (RT plus 24 months of ADT) and either the de-intensification arm (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies)

EXPLORATORY OBJECTIVES:

I. To compare changes in cardio-metabolic markers, including body mass index, and waist circumference, between the standard of care (RT plus 24 months of ADT) and either the de-intensification arm (RT plus 12 months of ADT) or intensification arm (RT plus 24 months of ADT plus apalutamide). (De-intensification and intensification studies) II. To develop a machine learning/artificial intelligence algorithm for radiotherapy quality assurance. (De-intensification and Intensification studies) III. To perform future translational correlative studies using biological and imaging data. (De-intensification and intensification studies) IV. Impact of position emission tomography (PET) use, measured by the proportion of times each type of imaging was used, in high-risk prostate cancer. (De-intensification and intensification studies)

PATIENT-REPORTED OUTCOMES OBJECTIVES:

PRIMARY OBJECTIVES:

I. To compare sexual and hormonal function related quality of life, as measured by the Expanded Prostate Cancer Index Composite-26 (EPIC), between the standard of care (RT plus 24 months of ADT) and the de-intensification arm (RT plus 12 months of ADT). (De-Intensification Study) II. To compare fatigue, as measured by the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue instrument, between the standard of care (RT plus 24 months of ADT) and the intensification arm (RT plus 24 months of ADT plus apalutamide). (Intensification Study)

SECONDARY OBJECTIVES:

I. To compare depression, as measured by the PROMIS-depression, between the standard of care (RT plus 24 months of ADT) and the de-intensification arm (RT plus 12 months of ADT). (De-Intensification Study) II. To compare depression, as measured by the PROMIS-depression, between the standard of care (RT plus 24 months of ADT) and the intensification arm (RT plus 24 months of ADT plus apalutamide). (Intensification Study)

EXPLORATORY OBJECTIVES:

I. To compare cognition, as measured by the Functional Assessment of Chronic Illness Therapy-Cognitive (FACT-Cog) perceived cognitive abilities subscale, between the standard of care (RT plus 24 months of ADT) and the de-intensification arm (RT plus 12 months of ADT). (De-Intensification Study) II. To compare bowel and urinary function related quality of life, as measured by the Expanded Prostate Cancer Index Composite-26 (EPIC), between the standard of care (RT plus 24 months of ADT) and the de-intensification arm (RT plus 12 months of ADT). (De-Intensification Study) III. To compare fatigue, as measured by the PROMIS-Fatigue instrument, between the standard of care (RT plus 24 months of ADT) and the de-intensification arm (RT plus 12 months of ADT). (De-Intensification Study) IV. To compare sexual and hormonal function related quality of life, as measured by the Expanded Prostate Cancer Index Composite-26 (EPIC), between the standard of care (RT plus 24 months of ADT) and the intensification arm (RT plus 24 months of ADT plus apalutamide). (Intensification Study) V. To compare bowel and urinary function related quality of life, as measured by the Expanded Prostate Cancer Index Composite-26 (EPIC), between the standard of care (RT plus 24 months of ADT) and the intensification arm (RT plus 24 months of ADT plus apalutamide). (Intensification Study) VI. To compare cognition, as measured by the Functional Assessment of Chronic Illness Therapy-Cognitive (FACT-Cog) perceived cognitive abilities subscale, between the standard of care (RT plus 24 months of ADT) and the intensification arm (RT plus 24 months of ADT plus apalutamide). (Intensification Study)

OUTLINE: Patients are randomized to 1 of 4 arms.

DE-INTENSIFICATION STUDY (DECIPHER SCORE =< 0.85):

ARM I: Patients undergo radiation therapy (RT) over 2-11 weeks and receive ADT (consisting of either leuprolide, goserelin, triptorelin, degarelix, buserelin, histrelin, or relugolix and bicalutamide or flutamide) for 24 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo RT over 2-11 weeks and receive ADT (consisting of either leuprolide, goserelin, triptorelin, degarelix, buserelin, histrelin, or relugolix and bicalutamide or flutamide) for 12 months in the absence of disease progression or unacceptable toxicity.

INTENSIFICATION STUDY (DECIPHER SCORE > 0.85 OR NODE POSITIVE):

ARM III: Patients undergo RT over 2-11 weeks and receive ADT (consisting of either leuprolide, goserelin, triptorelin, degarelix, buserelin, histrelin, or relugolix and bicalutamide or flutamide) for 24 months in the absence of disease progression or unacceptable toxicity.

ARM IV: Patients undergo RT over 2-11 weeks and receive ADT (consisting of either leuprolide, goserelin, triptorelin, degarelix, buserelin, histrelin, or relugolix) for 24 months in the absence of disease progression or unacceptable toxicity. Patients also receive apalutamide orally (PO) once daily (QD). Treatment repeats every 90 days for up to 8 cycles (24 months) in the absence of disease progression or unacceptable toxicity.

Patients undergo bone scan, positron emission tomography (PET) scan, computed tomography (CT) scan, and magnetic resonance imaging (MRI) at screening and as clinically indicated and may optionally undergo blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION
* Pathologically proven diagnosis of adenocarcinoma of prostate cancer within 180 days prior to registration
* High-risk disease defined as having at least one or more of the following:

  * PSA > 20 ng/mL prior to starting ADT

    * Note: Patients receiving a 5-alpha reductase inhibitor (ex. finasteride) at the time of enrollment are eligible. The baseline PSA value should be doubled for PSAs taken while on 5-alpha reductase inhibitors and the medication should be discontinued prior to randomization but a washout period is not required
  * cT3a-T4 by digital exam or imaging (American Joint Committee on Cancer [AJCC] 8th edition [Ed.])
  * Gleason score of 8-10
  * Node positive by conventional imaging with a short axis of at least 1.0 cm
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 120 days prior to registration;
  * Bone imaging within 120 days prior to registration;

    * Note: To be eligible, patient must have no definitive evidence of bone metastases (M0) on bone scan or sodium fluoride (NaF) PET within 120 days prior to registration (negative NaF PET/CT or negative Axumin or choline PET or negative fluciclovine, choline or prostate-specific membrane antigen (PSMA) PET within 120 days prior to registration is an acceptable substitute if they have been performed). Patients who have bone metastases established only fluciclovine, choline, or PSMA PET but not definitive on bone scan or NaF PET will still be eligible
  * CT or MRI of the pelvis within 120 days prior to registration (negative fluciclovine, choline, or PSMA PET within 120 days prior to registration is an acceptable substitute). As with bone staging, nodal staging for trial purposes will be based off of conventional imaging findings only
  * Patients with confirmed N1 metastases on conventional imaging (CT/MRI) as defined by >= 10 mm on short axis are eligible but will be automatically assigned to the intensification study. Patients who are positive by fluciclovine, choline, or PSMA PET (i.e. N1), but whose nodes do not meet traditional size criteria for positivity (i.e. they measure >= 10 mm on either the CT or MRI portion of the PET or on a dedicated CT or MRI) will not be considered N1 for the trial and will not automatically be assigned to the intensification study
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 120 days prior to registration
* Hemoglobin >= 9.0 g/dL, independent of transfusion and/or growth factors (within 120 days prior to registration)
* Platelet count >= 100 x 10^3/uL independent of transfusion and/or growth factors (within 120 days prior to registration)
* Creatinine clearance (CrCl) >= 30 mL/min estimated by Cockcroft-Gault equation (within 120 days prior to registration)

  * For Black patients whose renal function is not considered adequate by Cockcroft-Gault formula, an alternative formula that takes race into account (Chronic Kidney Disease Epidemiology Collaboration CKD-EPI formula) may be used for calculating creatinine clearance for trial eligibility
  * Either a CrCl >= 30 ml/min or calculated glomerular filtration rate (GFR) >= 30 will make a patient eligible
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 120 days prior to registration)

  * Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject is eligible
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (within 120 days prior to registration)
* Serum albumin >= 3.0 g/dL (within 120 days prior to registration)
* The patient must agree to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agree to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial and have a CD4 count >= 200 cells/microliter within 60 days prior to registration. Note: HIV testing is not required for eligibility for this protocol. Of note, for patients with HIV in the intensification trial randomized to apalutamide, highly active antiretroviral therapy (HAART) may need to be adjusted to medications that do not interact with apalutamide
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable after or on suppressive therapy within 60 days prior to registration, if indicated. Note: HBV viral testing is not required for eligibility for this protocol
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Note: Any patient with a cancer (other than keratinocyte carcinoma or carcinoma in situ or low-grade non-muscle invasive bladder cancer) who has been disease-free for less than 3 years must contact the principal investigator
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* PRIOR TO STEP 2 RANDOMIZATION
* Confirmation of Decipher score
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load within 60 days prior. Note: Apalutamide may interfere with HCV drugs. Patients on HCV medications should alert their infectious diseases physician if they get randomized to apalutamide due to the possibility that apalutamide can affect the bioavailability of some HCV medications. HCV viral testing is not required for eligibility for this protocol
* For patients entering the Intensification Cohort ONLY: Patients must discontinue or substitute concomitant medications known to lower the seizure threshold at least 30 days prior to Step 2 randomization

Exclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION:
* Definitive radiologic evidence of metastatic disease outside of the pelvic nodes (M1a, M1b or M1c) on conventional imaging (i.e. bone scan, CT scan, MRI)
* Prior systemic chemotherapy within =< 3 years prior to registration; note that prior chemotherapy for a different cancer is allowed (completed > 3 years prior to registration
* Prior radical prostatectomy
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Current use of 5-alpha reductase inhibitor. NOTE: If the alpha reductase inhibitor is stopped prior to randomization the patient is eligible
* History of any of the following:

  * Seizure disorder
  * Current severe or unstable angina
  * New York Heart Association Functional Classification III/IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
  * History of any condition that in the opinion of the investigator, would preclude participation in this study
* Evidence of any of the following at registration:

  * Active uncontrolled infection requiring IV antibiotics
  * Baseline severe hepatic impairment (Child Pugh Class C)
  * Inability to swallow oral pills
  * Any current condition that in the opinion of the investigator, would preclude participation in this study
* Prior pharmacologic androgen ablation for prostate cancer is allowed only if the onset of androgen ablation (both luteinizing hormone-releasing hormone [LHRH] agonist and oral anti-androgen) is =< 60 days prior to registration; Please note: baseline PSA must be obtained prior to the start of any ADT
* PRIOR TO STEP 2 RANDOMIZATION:
* Evidence of known gastrointestinal disorder affecting absorption of oral medications at registration
* For patients entering the Intensification Cohort ONLY: Presence of uncontrolled hypertension (persistent systolic blood pressure [BP] >= 160 mmHg or diastolic BP >= 100 mmHg). Subjects with a history of hypertension are allowed, provided that BP is controlled to within these limits by anti-hypertensive treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2753 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival (MFS) | From randomization to the date of detection of distant metastasis on standard imaging or date of death from any cause, assessed up to 13 years
  Assessed based on conventional imaging. MFS will be estimated using the Kaplan-Meier method (Kaplan 1958).
Sexual quality of life (De-intensification study) | Up to 13 years
  Measured by Expanded Prostate Cancer Index Composite-26 sexual domain
Hormonal quality of life (De-intensification study) | Up to 13 years
  Measured by EPIC-26 hormonal domain
Fatigue (Intensification study) | Up to 13 years
  Measured by Patient Reported Outcomes Measurement Information Systems (PROMIS) Fatigue short form (SF)

SECONDARY OUTCOMES:
MFS | From randomization to the date of detection of distant metastasis on standard imaging or date of death from any cause, assessed up to 13 years
  Assessed based on standard or molecular, if available, imaging. MFS will be estimated using the Kaplan-Meier method (Kaplan 1958)
Overall survival | From the date of randomization to the date of death or last known follow-up date, with patients alive at the last known follow-up time treated as censored, assessed up to 13 years
  Will be estimated using the Kaplan-Meier method and treatment arms compared using the stratified log-rank test (Kaplan 1958).
Prostate cancer specific mortality (PCSM) | From the date of randomization to the date of prostate cancer death, assessed up to 13 years
Prostate specific antigen (PSA) failure-free survival with non-castrate testosterone and no additional therapies | From the date of randomization to the date event, or death or censored at the last known follow-up date, assessed up to 13 years
  PSA failure-free survival will be estimated using the Kaplan-Meier method and treatment arms compared using the stratified log-rank test (Kaplan 1958).
Time to testosterone recovery | Up to 13 years
  Defined as testosterone that is non-castrate.
Time to PSA failure or salvage therapy | Up to 13 years
Testosterone levels at the time of PSA failure and metastases | Up to 13 years
Incidence of adverse events | Up to 13 years
  Measured by the Common Terminology Criteria for Adverse Events (CTCAE ) version (v) 5.0 and Patient Reported Outcomes (PRO)-CTCAE.
Depression (De-intensification study) | Up to 13 years
  Measured by the PROMIS Depression
Depression (Intensification study) | Up to 13 years
  Measured by the PROMIS Depression

OTHER OUTCOMES:
Cardio-metabolic markers including body mass index and waist circumference | Up to 13 years
Machine learning/artificial intelligence algorithm | Up to 13 years
Impact of PET use | Up to 13 years
  Measured by the proportion of times each type of imaging was used.
Fatigue (De-intensification study) | Up to 13 years
  Measured by PROMIS- Fatigue Short Form (SF)
Bowel and urinary quality of life (De-intensification study) | Up to 13 years
  Measured by EPIC-26 bowel and urinary domains.
Cognition (De-intensification study) | Up to 13 years
  Measured by the Functional Assessment of Chronic Illness Therapy-Cognition (FACIT-Cog) perceived cognitive abilities subscale.
Sexual, hormonal, bowel, and urinary quality of life (Intensification study) | Up to 13 years
  Measured by EPIC-26
Cognition (Intensification study) | Up to 13 years
  Measured by the FACIT-Cog perceived cognitive abilities subscale.
Primary outcome treatment effect by sex | Up to 13 years
  Estimates of the primary outcome treatment effect and the corresponding 95% confidence intervals (CIs) by sex.
Primary outcome treatment effect by race | Up to 13 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by race.
Primary outcome treatment effect by ethnicity | Up to 13 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Nguyen, Principal Investigator — NRG Oncology
Locations (602):
- United States (594):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Phoenix, Phoenix, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Enloe Medical Center, Chico, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin General Hospital, Greenbrae, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Providence Queen of The Valley, Napa, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - California Protons Cancer Therapy Center, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - UCSF Cancer Center - San Mateo, San Mateo, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - City of Hope South Bay, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - GenesisCare USA - Lakewood Ranch, Lakewood Rch, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Miami Cancer Institute at Plantation, Plantation, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Alton Memorial Hospital, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Saint Joseph Hospital East, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Veterans Administration Medical Center-Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Capital Region Medical Center, Largo, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Clara Maass Medical Center, Belleville, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Northwell Health Physicians Partners Radiation Medicine at Queens, Forest Hills, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Queens Cancer Center, Rego Park, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - UNC Health Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - UNC Health Cancer Care Wakefield, Raleigh, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Yolanda G Barco Oncology Institute, Meadville, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital-Quakertown Campus, Quakertown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC Health Florence Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Beaufort Memorial/New River Cancer Center, Okatie, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Oncology Group-Maryville, Maryville, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (8):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan